CLINICAL TRIAL: NCT00352703
Title: An Open-label, Single-arm Study of Palifermin for Reduction of Mucositis in Subjects With Non-Hodgkin's Lymphoma or Multiple Myeloma Undergoing High-Dose Chemotherapy and Autologous Peripheral Blood Stem Cell (PBSC) Transplantation
Brief Title: PROMPT - Palifermin in Reduction of Oral Mucositis in PBSC Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20050100
Record Dates: First submitted 2006-07-13; First posted 2006-07-17 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Non-Hodgkin's Lymphoma; Multiple Myeloma
Keywords: Oral mucositis; Non-Hodgkin's lymphoma (NHL); conditioning chemotherapy; autologous PBSCT; multiple myeloma (MM); Melphalan
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma; Stomatitis | interventions — Fibroblast Growth Factor 7

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kepivance (palifermin) 60 μg/kg/day IV (Experimental): 60 μg/kg/day IV for 3 consecutive days before the conditioning regimen and 3 consecutive days after the peripheral blood stem cell transplantation.
  Interventions: Drug: Kepivance (Palifermin)

INTERVENTIONS:
Drug: Kepivance (Palifermin)

SUMMARY:
This is an open-label, single-arm, multicentre study conducted in Spain to estimate the effectiveness of palifermin administered at a dose of 60 mg/kg/day IV for 3 consecutive days before the start of the conditioning regimen and for 3 consecutive days after autologous PBSCT for treating oral mucositis in patients with NHL and MM who have received high-dose conditioning chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Non-Hodgkin's lymphoma (NHL) subjects scheduled to receive BEAM conditioning chemotherapy followed by autologous PBSCT, or multiple myeloma (MM) subjects scheduled to receive high-dose Melphalan (200 mg/m2) conditioning chemotherapy, in a one or two-day schedule, followed by autologous PBSCT
* ≥Age 18 years
* ECOG performance status <= 2. In the MM group, ECOG status >2 will be accepted provided that it is exclusively due to MM (e.g. pathological fracture)
* Adequate pulmonary function as measured by a corrected carbon monoxide (CO) diffusing capacity (DLCO) ≥ 60% of predicted
* Left ventricular ejection fraction (LVEF) ≥ 50%
* Minimum of 1.5 x 10^6 CD34+ cells/kg for autologous transplantation
* Adequate haematological function (ANC ≥ 1.5 x 10^9/L and platelet count ≥ 100 x 10^9/L)
* Serum creatinine <= 2.0 mg/dL
* Total bilirubin <= 2 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 4.0 x IULN
* Negative serum or urine pregnancy test for women of child bearing potential within 14 days prior to enrolment
* Each subject must give informed consent directly or through a legally acceptable representative before participating in any study specific procedure, or receiving any study medication. Exclusion Criteria:
* History of or concurrent cancer other than NHL or MM
* Prior treatment with palifermin, or other keratinocyte growth factors (eg, KGF-2)- Prior autologous or allogeneic transplants
* Oral abnormalities defined as baseline oral assessment of WHO grade >0
* Other investigational procedures are excluded
* Subject currently is enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study(s), or subject is receiving other investigational agent(s)
* Subject of child-bearing potential is evidently pregnant (eg, positive HCG test) or is breast feeding
* Subject is not using adequate contraceptive precautions
* Known to be sero-positive for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV)
* Subject has known sensitivity to any of the products to be administered during dosing, including E coli-derived products
* Subject has previously been treated on this study or with other keratinocyte growth factors
* Unwilling or unable to complete the patient-reported outcome questionnaires
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2006-04; Primary Completion 2007-04 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoints are the incidence (%) and duration of severe oral mucositis (WHO grades 3 or 4). | Up to 40 days
  The study consisted of a screening period of up to 42 days to determine subject eligibility, followed by a treatment period of a maximum of 40 days.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Biovitrum AB

REFERENCES:
- See also: FDA-approved Drug Labeling — http://www.kepivance.com/